CLINICAL TRIAL: NCT01984983
Title: A Phase I, Randomized, Observer-blind, Placebo Controlled Study to Assess the Safety, Reactogenicity, and Immunogenicity of a Venezuelan Equine Encephalitis DNA Vaccine Candidate Administered Intramuscularly or Intradermally by Electroporation to Healthy Adults
Brief Title: Study of a DNA-based Venezuelan Equine Encephalitis Virus DNA Vaccine Administered by Electroporation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ichor Medical Systems Incorporated (Industry)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMS-VEEV-001
Record Dates: First submitted 2013-09-23; First posted 2013-11-15 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Venezuelan Equine Encephalitis Virus Infection
Keywords: Venezuelan equine encephalitis virus; DNA vaccine; electroporation; intradermal; intramuscular
MeSH Terms: conditions — Encephalomyelitis, Venezuelan Equine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- VEEV DNA Vaccine 0.5 mg/ml Intramuscular (Experimental): Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
  Interventions: Biological: Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
- VEEV DNA Vaccine 0.5 mg/ml Intradermal (Experimental): Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
  Interventions: Biological: Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
- VEEV DNA Vaccine 2.0 mg/ml Intramuscular (Experimental): Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
  Interventions: Biological: Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
- VEEV DNA Vaccine 2.0 mg/ml Intradermal (Experimental): Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
  Interventions: Biological: Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
- Placebo: 0.9% saline (Placebo Comparator): 0.9% saline
  Interventions: Other: 0.9% saline placebo

INTERVENTIONS:
Biological: Venezuelan Equine Encephalitis Virus DNA Vaccine Candidate
  Arms: VEEV DNA Vaccine 0.5 mg/ml Intradermal; VEEV DNA Vaccine 0.5 mg/ml Intramuscular; VEEV DNA Vaccine 2.0 mg/ml Intradermal; VEEV DNA Vaccine 2.0 mg/ml Intramuscular
Other: 0.9% saline placebo
  Arms: Placebo: 0.9% saline

SUMMARY:
The Phase I study will assess the basic safety, tolerability, and immunogenicity of a DNA-based Venezuelan equine encephalitis virus (VEEV)vaccine candidate delivered by electroporation . The study will enroll 40 healthy adult volunteers ages 18-49 and will comprise evaluation of intradermal or intramuscular administration by electroporation. Administration of the vaccine candidate will be at two DNA dose levels (0.5 mg/ml and 2.0 mg/ml) for each route of administration. Electroporation will be administered using the TriGrid Delivery System devices for intramuscular and intradermal delivery. An additional group of subjects will serve as a placebo control, receiving injections of saline with electroporation. The overall goal of this study will be to determine if further human clinical studies of the vaccine candidate are warranted and, if so, to aid in the selection of dose and route of administration for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or non-pregnant, non-lactating female, ages 18-49 (inclusive) at time of screening
* Have provided written informed consent before screening
* Free of clinically significant health problems or clinical lab abnormalities, as determined by pertinent medical history, lab evaluations, and clinical examination before entry into the study
* Available and able to participate for all study visits and procedures
* If sexually active, known to be at least 1 year post-menopausal, or willing to use an effective method of contraception (e.g., birth control pill, diaphragm, cervical cap, intrauterine device, condom, anatomical sterility [self or partner]) from the date of screening until at least 6 months after the last injection
* Negative VEEV IgG antibody test result at screening (ELISA)

Exclusion Criteria:

* History or serologic evidence of prior infection with VEE virus or prior participation in a VEE virus vaccine trial
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
* History of Guillain-Barre Syndrome
* Ongoing participation in another clinical trial
* Receipt or planned receipt of any experimental or licensed vaccine, except for a licensed seasonal influenza vaccine, within the period 30 days prior to initial injection through 60 days after the Day 70 follow-up. (~ 6 month period in total)
* Receipt or planned receipt of any allergy treatments involving antigen injections within the period 30 days prior to the first injection through the period 60 days after Study Day 70 (~6 month period in total)
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for the eligible injection sites (left and right medial deltoid region) exceeds 40 mm
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
* Therapeutic or traumatic metal implant in the skin or muscle of either deltoid region.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, EKG, and/or laboratory screening test
* Pregnant or lactating female, or female who intends to become pregnant during the study period
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection
* Administration of chronic (defined as more than 14 days) immunosuppressant's or other immune-modifying drugs within 6 months of study entry
* For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day; Inhaled and topical steroids are allowed
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child
* Syncopal episode within 12 months of screening
* Suspected or known current alcohol abuse as defined by the American Psychiatric Association in DSM IV (Diagnostic and Statistical Manual of Mental Disorders-4th edition)
* Chronic or active illicit and/or intravenous drug use by history
* Unwilling to allow storage and use of blood for future alphavirus-related research
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The nature, frequency, and severity of local and systemic adverse events or serious adverse events associated with electroporation-based administration of the VEEV DNA vaccine candidate | 12 months

SECONDARY OUTCOMES:
The frequency, magnitude, and duration of serum anti-VEEV antibody responses | 12 months
  Anti-VEEV immune response will be assessed by 80% Plaque Reducing Neutralization Test (PRNT80). PRNT80 titers of >= 1:10 will constitute a response.
Response to a questionnaire based assessment of acute procedure tolerability. | 8 weeks
  Immediately following procedure administration, subjects will complete a Visual Analog Scale (VAS) based questionnaire to assess procedure tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Accelovance, San Diego, California, United States

REFERENCES:
- [Derived] Hannaman D, Dupuy LC, Ellefsen B, Schmaljohn CS. A Phase 1 clinical trial of a DNA vaccine for Venezuelan equine encephalitis delivered by intramuscular or intradermal electroporation. Vaccine. 2016 Jun 30;34(31):3607-12. doi: 10.1016/j.vaccine.2016.04.077. Epub 2016 May 17. PMID 27206386